CLINICAL TRIAL: NCT04656119
Title: Discovery of Biomarkers Related to the Efficacy and Adverse Reactions of Immune Checkpoint Inhibitors Based on Metabolism-genomics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Lihong Liu, Director of Pharmacy department, Beijing Chao Yang Hospital
Other Study IDs: 2020-K-508
Record Dates: First submitted 2020-11-18; First posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-11

CONDITIONS: Cancer
Keywords: Immune checkpoint inhibitors; Immune-related adverse events; Genomics; Metabonomics
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients without irAEs or patients with good efficacy
  Interventions: Other: there is no intervention in our study
- patients with irAEs or patients with poor efficacy
  Interventions: Other: there is no intervention in our study

INTERVENTIONS:
Other: there is no intervention in our study — there is no intervention in our study

SUMMARY:
Immune checkpoint inhibitors (ICIs) are an important breakthrough in cancer therapy and have been increasingly used.However, ICIs can cause a unique spectrum of side effects termed immune-related adverse events (irAEs),which can affect any organ systems and in some cases are fulminant or even fatal.In clinical practice, irAEs and clinical efficacy maybe various for patients with same standard treatment, and some studies have shown that gene and metabolic differences in cancer patients may be an important factor. In this project, peripheral blood samples from cancer patients will be collected prospectively at baseline, and at regular intervals (2 cycles, about 6 weeks) for about 30 weeks, then these blood samples will be analyzed using the technique of genomics, metabonomics.

The investigators aim to find biomarkers associated with irAE or clinical efficacy. When the sample size and data is big enough, the investigators plan to establish a prediction model using machine learning to access the safety and efficacy of ICIs for cancer patients. Our study have important clinical implications in the prediction and early management of severe, potentially life-threatening immune-related toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant tumor, no relative contraindications for immunotherapy, in line with the standards of immunotherapy
* Receive immune checkpoint inhibitors (ICIs) for the first time or have received ICIs but no immune-related adverse reactions have occurred
* Have provided informed consent, are willing to participate in study and routine follow-up
* At least one measurable lesion according to Guidelines for response criteria for use in trials testing immunotherapeutics (iRECIST)

Exclusion Criteria:

* Active, known, suspected or a documented history of autoimmune disease
* Eastern Cooperative Oncology Group(ECOG) performance status 3-4
* Long-term hormone therapy，corticosteroids (>10mg/day prednisone curative dose)
* Subjects with human immunodeficiency virus (HIV)
* Subjects with other tumors
* Myocardial infarction, poorly control led arrhythmia, New York Heart Association (NYHA) standard III-IV cardiac insufficiency or left ventricular ejection fraction (LVEF)<50% in the last 6 month
* Active tuberculosis
* Active or a documented history of interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severely impaired lung function
* Common Terminology Criteria for Adverse Events (CTCAE) peripheral neuropathy grade≥2
* History of alcohol abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the participants make up the study population
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-11-03 (Actual); Primary Completion 2022-11-03 (Estimated); Study Completion 2025-11-03 (Estimated)

PRIMARY OUTCOMES:
immune-related adverse events incidence | November,2020-November,2025

SECONDARY OUTCOMES:
Complete response (CR) | November,2020-November,2025
Partial response (PR) | November,2020-November,2025
Stable disease (SD) | November,2020-November,2025
Progressive disease (PD) | November,2020-November,2025

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chao-yang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No